CLINICAL TRIAL: NCT06114979
Title: Silodosin vs Placebo in the Treatment of Female Lower Urinary Tract Symptoms: A Randomized Controlled Trial
Brief Title: Silodosin vs Placebo in the Treatment of Female LUTS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Collaborators: Amiri Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Silodosin for female LUTS; 937/2018 (Registry Identifier: Research Coordination Committee)
Record Dates: First submitted 2023-10-20; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Silodosin; LUTS; Female
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — silodosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silodosin (Active Comparator): Patients will receive 8 mg of Silodosin tablet once daily.
  Interventions: Drug: Silodosin
- Placebo (Placebo Comparator): Patients will receive placebo pill once daily,
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silodosin — Each patient will receive 8 mg of silodosin tablet once daily.
  Arms: Silodosin
Drug: Placebo — Each patient will receive placebo tablet.
  Arms: Placebo

SUMMARY:
This trial will be conducted to study the efficacy and safety of Silodosin in the treatment of female lower urinary tract symptoms.

DETAILED DESCRIPTION:
The double blinded randomized controlled trial will evaluate efficacy and safety of silodosin in treatment of female lower urinary tract symptoms by comparing with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Females complaining of lower urinary tract symptoms
* IPSS ≥ 8 or OAB - V8 score ≥ 8

Exclusion Criteria:

1. Patients with documented hypersensitivity to Silodosin.
2. Patients receiving alpha blockers or anticholinergic medications for any other reason.
3. Patients with history of orthostatic hypotension.
4. Pregnant or breastfeeding females.
5. Patients with stress urinary incontinence.
6. Patients with active urinary tract infection.
7. History of previous pelvic surgery or radiation.
8. Patient with diabetes mellitus.
9. Patients diagnosed with bladder cancer.
10. Patients with hepatic impairment (Child-Pugh score >9).
11. Patients with severe renal impairment with creatinine clearance of less than 10 mL/min.
12. Patients planned to undergo any ophthalmic procedure.
13. Patients with history of urinary retention or gastric retention.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 278 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score | 8 weeks
  International Prostate Symptom Score will be recorded for each patient. The score ranged between 7 and 35. Higher scores means worse outcome.
Overactive Bladder Validated 8-question | 8 weeks
  Overactive Bladder Validated 8-question will be recorded for each patient. The score ranged between 2 and 42. Higher scores means worse outcome.

SECONDARY OUTCOMES:
Uroflometry | 8 weeks
  Voided volume , Maximum flow, Voiding time, Post void residual
Adverse events | 8 weeks
  Side effects of the treatment will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Tariq F AL-Shaiji, MD, Principal Investigator — Amiri Hospital

IPD SHARING:
Plan to Share IPD: No